CLINICAL TRIAL: NCT04500678
Title: A 72 Week, Randomized, Open-label vs Observation Study to Assess the Potential Immuno-virologic Benefit of Metformin in HIV-infected Individuals Receiving Antiretroviral Therapy
Brief Title: Impact of Metformin on Immuno-virologic Parameters in HIV
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Hawaii (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Cecilia Shikuma, Professor, Medicine, University of Hawaii
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: H046
Record Dates: First submitted 2020-07-31; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Metformin vs Observation
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin (Experimental): Metformin 500 mg Extended Release (ER) qd increasing to 1000 mg ER qd at week 4 and continued to week 48.
  Interventions: Drug: Metformin
- Observation (No Intervention): Observed without metformin

INTERVENTIONS:
Drug: Metformin — Metformin 500 mg Extended Release (ER) qd increasing to 1000 mg ER qd at week 4 and continued to week 48.
  Arms: Metformin

SUMMARY:
Non-diabetic, aviremic HIV-infected individuals on antiretroviral therapy (ART) will be randomized to metformin therapy or to observation for 72 weeks. Primary objective is to assess change over 72 weeks in CD4 T cell negative checkpoint receptors (PD-1 and TIGIT). As secondary objectives the study will look at 72 week change in other immuno-virologic parameters (CD8 T cell negative checkpoint receptors, plasma indoleamine 2,3-dioxygenase (IDO) levels and CD4 T cell and monocyte intracellular HIV DNA and HIV RNA. The study will also explore the 72 week impact of metformin on change in carotid intima-media thickness (cIMT) as a surrogate marker of atherosclerosis, on neuropsychological (NP) performance, strength, and change in body composition.

ELIGIBILITY:
Inclusion Criteria:

* HIV+
* On suppressive ART stable for > 1 year
* Plasma HIV RNA < 50 copies/mL within 3 months of entry, with no HIV RNA > 200 copies/mL within the past 6 months prior to entry
* Age >40 years
* Ability and willingness to provide written informed consent

Exclusion Criteria:

* Uncontrolled chronic medical condition or cancer
* Acute illness within 2 weeks of entry
* Diagnosis of diabetes by history, fasting blood glucose >126, or by HgbA1c > 6.5
* Chronic, uncontrolled diarrhea
* Known hypersensitivity or contraindication to metformin use
* Current presence of hepatitis C including currently on or intent to start therapy for hepatitis C within the 48 week duration of study.
* Serum B12 level below the reference normal range as listed by the commercial lab utilized for this study (Diagnostic Laboratory Services)
* Pregnancy, or intent to become pregnant or nursing an infant
* Any immunomodulator, HIV vaccine, any other vaccine, or investigational therapy within 30 days of study entry.
* Current uncontrolled coronary artery disease or NYHA Class 3 or 4 congestive heart failure
* History of liver cirrhosis
* Current use of zidovudine, stavudine or didanosine
* The following lab values

  * Hemoglobin < 9.0 g/dL
  * Absolute neutrophil count < 1000/μL
  * Platelet count < 50,000/μL
  * AST (SGOT) and ALT (SGPT) > 5x upper limit of normal (ULN)
  * Calculated creatinine clearance (Cockcroft and Gault) < 50 ml/min
* Active or recent past history (within past 2 years) of illicit substance or alcohol use or abuse which, in the judgment of the Investigator, will interfere with the patient's ability to comply with the protocol requirements
* Patients, who, in the opinion of the Investigator, are unable to comply with the dosing schedule and protocol evaluation or for whom the study may not be advisable

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
CD4 T cell PD1+TIGIT+ | Entry to week 72
  Comparison of change over time in percentage of CD4 T cells bearing the PD1+TIGIT+ surface markers in peripheral blood mononuclear cells (PBMC) in the treatment (metformin) arm compared to the observation arm

SECONDARY OUTCOMES:
CD8 T cell PD1+TIGIT+ | Entry to week 72
  Comparison of change over time in percentage of CD8 T cells bearing the PD1+TIGIT+ surface markers in PBMCs in the 2 study arms
Plasma levels of indoleamine 2,3-dioxygenase (IDO) | Entry to week 72
  Comparison of change over time in the levels of IDO [assessed as a ratio of L-kynurenine (kyn) to substrate tryptophan (trp)] in mass spectrometry assays
Peripheral blood CD4 T cell intracellular HIV DNA | Entry to week 72
  Comparison of change over time in the number of intracellular HIV DNA copies per million CD4 T cells in PBMC in the 2 study arms
Peripheral blood CD4 T cell intracellular HIV RNA | Entry to week 72
  Comparison of change over time in the number of intracellular HIV RNA copies per million CD4 T cells in PBMC in the 2 study arms
Peripheral blood monocyte intracellular HIV DNA | Entry to week 72
  Comparison of change over time in the number of intracellular HIV DNA copies per million monocytes in PBMC in the 2 study arms
Peripheral blood monocyte intracellular HIV RNA | Entry to week 72
  Comparison of change over time in the number of intracellular HIV RNA copies per million monocytes in PBMC in the 2 study arms

OTHER OUTCOMES:
Safety and Tolerability: # of grade 2 or greater adverse events in each arm | Entry to week 72
  Comparison of the # of grade 2 or greater adverse events in the 2 arms
Carotid intima-media thickness | Entry to week 72
  Comparison of change over time in the thickness of the right carotid intima-media thickness (mm) as assessed by carotid ultrasound in the 2 study arms
Neuropsychological testing global Z score | Entry to week 72
  Comparison of change over time in the age, gender and education-adjusted neuropsychological testing global Z score in the 2 study arms [The z score has a mean of zero and a standard deviation of 1; higher than 0 is better cognitive performance and lower than 0 is lower performance than the mean]
Beck's Depression Index II score | Entry to week 72
  Comparison of change over time in the Beck's Depression Index II score in the 2 study arms [21-item rating scale with maximum score of 63; higher scores are indicative of worse depression]
Handgrip | Entry to week 72
  Comparison of change over time in handgrip strength (kg) as assessed by a handgrip dynamometer in the 2 study arms
Total lean tissue by dual energy absorptiometry (DXA) | Entry to week 72
  Comparison of change over time in total lean tissue (kg) as assessed by DXA in the 2 study arms

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia M Shikuma, MD, Principal Investigator — University of Hawaii
Locations (1):
- John A. Burns School of Medicine, University of Hawaii - Manoa, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: Yes
Dataset will be available to other researchers upon request once the primary manuscript is written
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the study analyses are completed and primary manuscript is published, and for a duration of at least 5 years afterwards
Access Criteria: De-identified dataset will be provided upon request to legitimate researchers